CLINICAL TRIAL: NCT05562219
Title: A Randomized, Double-Masked, Placebo-Controlled, Multicenter, Phase II Clinical Study of the Efficacy and Safety of QA108 Granules in the Treatment of Intermediate Age-Related Macular Degeneration
Brief Title: QA108 Phase II Study in Subjects With Intermediate Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Smilebiotek Zhuhai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QA108
Record Dates: First submitted 2022-09-13; First posted 2022-09-30 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Intermediate Age-Related Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group(QA108 granules) (Experimental): QA108 granules, 7.5 g/bag,2 bags/time, BID
  Interventions: Drug: QA108 granules
- Placebo group(QA108 granule simulants) (Placebo Comparator): QA108 granule simulants, 7.5 g/bag,2 bags/time, BID
  Interventions: Drug: QA108 granules placebo

INTERVENTIONS:
Drug: QA108 granules — Take the medication as required for 24 weeks
  Arms: Treatment group(QA108 granules)
Drug: QA108 granules placebo — Take the medication as required for 24 weeks
  Arms: Placebo group(QA108 granule simulants)

SUMMARY:
This is a phase 2, randomized, double-masked, placebo-controlled, multicenter study. To evaluate the efficacy and safety of QA108 granules in the treatment of intermediate age-related macular degeneration.

DETAILED DESCRIPTION:
Approximately 12 sites will randomize a total of approximately 120 subjects . The subject randomization code table is generated using block randomization. Randomization of not less than 120 cases receiving treatment (treatment and placebo groups) at a ratio of 1:1 for the treatment and control groups.

Clinic study visits will occur on Day -7 to Day -1(Screening/Baseline)(Randomization); Treatment Visits for weeks 4, 8, 12,16,20,and 24 (all ± 3 days); sites will contact each subject to update efficacy date and adverse events (AEs) and review concomitant medications (CMs).

ELIGIBILITY:
Inclusion Criteria:

1. The study eye is diagnosed by western medicine with intermediate age-related macular degeneration, i.e., at least one large drusen (≥ 125 μm in diameter) is visible within two papillary diameters (PD) away from the fovea;
2. Consistent with the TCM diagnosis of type of Yang-hyperactivity due to Yin-deficiency;
3. Age 45 to 85 years old (both inclusive), male or female;
4. The study eye has a BCVA of 83-34 ETDRS letters (inclusive), which is equivalent to a Snellen visual acuity of 20/25 to 20/200 (inclusive);
5. The subject is voluntary to participate in this clinical study, provide informed consent, and sign the informed consent form.

Exclusion Criteria:

1. The study eye is with concomitant eye disorders that may interfere with the observation of the trial as judged by the investigator, including pathological myopia, glaucoma, diabetic retinopathy, retinal vein occlusion, uveitis, retinal detachment, optic neuropathy (optic neuritis, atrophy, papilledema), and macular hole;
2. The study eye has an intraocular pressure (IOP) ≥ 25 mmHg;
3. The study eye is presented with GA;
4. Previous ophthalmic surgery in the study eye: vitrectomy, macular translocation;
5. Aphakia (except pseudophakia) or posterior capsule rupture (except YAG laser posterior capsulotomy after IOL implantation at more than 1 month prior to screening) of the study eye;
6. Any intraocular or periocular surgery of the study eye and intraocular surgery (except eyelid surgery) of the non-study eye within 3 months;
7. The study eye is diagnosed with cataract affecting fundus observation, which may require cataract surgery within 6 months at the discretion of the investigator;
8. The study eye has received the following treatment within 3 months prior to screening: macular laser photocoagulation and micro-pulse laser therapy;
9. The patient received relevant TCM treatment within 1 month prior to screening;
10. Active ocular infection in either eye;
11. The non-study eye has a BCVA of less than 19 ETDRS letters (not inclusive);
12. Known allergy to the therapeutic or diagnostic drug used in the study protocol, including the single drug components in the study drugs;
13. Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg after regular use of antihypertensive drugs);
14. Patients with platelet count ≤ 100 × 109/L, total bilirubin (TBIL) > upper limit of normal (ULN), alanine transaminase (ALT) or aspartate aminotransferase (AST) > 1.5 × ULN, and blood creatinine > ULN;
15. Pregnant women, women who are breastfeeding, those who plan for pregnancy in the next six months, or those who are unwilling to take effective birth controls during the study course and until six months after drug withdrawal;
16. Any uncontrollable clinical disorder prior to the start of treatment, such as severe psychiatric, neurological, respiratory, immunological, hematological, and cardiac system diseases, and malignant tumors;
17. Subjects who have participated in other clinical trials within 3 months prior to this trial;
18. Patients who are unsuitable for participating at the discretion of the investigator.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in drusen area . | weeks 24
  1. change from baseline in drusen area as measured by optical coherence tomography (OCT)
  2. assessments will be conducted by the central reading center (CRC)

SECONDARY OUTCOMES:
Percentage change from baseline in drusen area | weeks 4,8,12,16,20
  change from baseline in drusen area as measured by optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital (PUMCH), Beijing, China